CLINICAL TRIAL: NCT04242368
Title: Hypertonic Versus Isotonic Saline Irrigations for Chronic Rhinosinusitis
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: COVID-19 pandemic, unable to recruit and conduct study procedures per state, local, and university policies.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Neelaysh Vukkadala, Resident Physician, Department of Otolaryngology - Head and Neck Surgery, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-53836
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
Keywords: chronic rhinosinusitis; nasal rinses; nasal irrigations
MeSH Terms: conditions — Disease | interventions — Sodium Chloride; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Isotonic rinse, then hypertonic rinse (Active Comparator): Participants will start with a one week washout period without rinses. Then they will complete twice daily sinus rinses isotonic saline for two weeks. Next they will have a one week washout period without rinses. Then they will cross-over and complete hypertonic saline sinus rinses for two weeks. Participants will maintain fluticasone treatment throughout the study.
  Interventions: Drug: Isotonic saline; Drug: Hypertonic Nasal Wash; Drug: Fluticasone Propionate
- Hypertonic rinse, then isotonic rinse (Experimental): Participants will start with a one week washout period without rinses. Then they will complete twice daily sinus rinses of hypertonic saline for two weeks. Next they will have a one week washout period without rinses. Then they will cross-over and complete isotonic saline sinus rinses for two weeks. Participants will maintain fluticasone treatment throughout the study.
  Fluticasone propionate nasal spray - two sprays to each nare twice a day used for the entire study duration
  Interventions: Drug: Isotonic saline; Drug: Hypertonic Nasal Wash; Drug: Fluticasone Propionate

INTERVENTIONS:
Drug: Isotonic saline — Nasal isotonic saline irrigation (240 mL, 0.9% NaCl) administered through nasal rinse bottle.
Drug: Hypertonic Nasal Wash — Nasal hypertonic saline irrigation (240 mL, 1.8% NaCl) administered through nasal rinse bottle.
Drug: Fluticasone Propionate — Fluticasone nasal spray administered two sprays to each nare twice a day
  Other Names: Flonase

SUMMARY:
The study aims to determine the safety and efficacy of buffered hypertonic (1.8%) saline nasal rinses as compared to isotonic saline nasal rinses in patients with chronic rhinosinusitis (CRS). Evidence from basic science research suggests that hypertonic solutions may have beneficial effects over isotonic saline rinses; however prior clinical studies on this topic have been inconclusive and limited due to highly variable inclusion criteria, large variability in the volume and concentration of irrigation solution, and inconsistent outcome measures. The goal of the study is to utilize a cross over study design to directly compare the impact of two different types of saline irrigation.

Primary aim:

Compare the efficacy of buffered hypertonic saline irrigations to buffered isotonic saline irrigations on patient reported outcome measures of chronic rhinosinusitis symptoms and nasal obstruction in patients with CRS. Based on in vivo data and prior clinical studies, the investigators expect participants will experience greater symptom improvement with hypertonic saline rinses as compared to isotonic saline irrigations.

Hypothesis: Participants will have greater improvement in patient reported outcome measures (SNOT-22 and NOSE) when using buffered hypertonic sinus irrigations as compared to buffered isotonic saline irrigations.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of chronic rhinosinusitis with or without polyposis based on the criteria outlined in the American Academy of Otolaryngology-Head and Neck Surgery's Clinical Practice Guideline
2. SNOT-22 score >/= 20

Exclusion Criteria:

1. Sinus surgery within 30 days of beginning the study
2. Oral steroid use within two weeks of study initiation
3. Active sinus exacerbation or sinus exacerbation within two weeks of starting the study
4. Allergies or contraindications to fluticasone nasal spray

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Mean change in SNOT-22 score | Beginning of week 2 and end of week 3 of the respective treatment period
  Participants will complete the Sinonasal Outcome Test (SNOT)-22, a validated questionnaire for assessing symptoms of chronic rhinosinusitis, before and after completing each intervention.
  SNOT-22 is a validated scale which measures sinonasal symptoms for sinusitis patients. The 22 questions are rated on a scale of 0-5 for a maximum total score of 110. Higher scores represent more symptomatic patients.
Mean change in NOSE score | Beginning of week 2 and end of week 3 of the respective treatment period
  Participants will complete the Nasal Obstruction Symptom Evaluation (NOSE), a validated questionnaire for assessing symptoms of nasal obstruction, before and after completing each intervention.
  NOSE scores can range from 5 to 100, with higher scores indicating worse symptoms. Classes are mild (5-25), moderate (30-50), severe (55-75), and severe (80-100).

SECONDARY OUTCOMES:
Participant-reported compliance with sinus rinses | From the beginning of week 2 to the end of week 3 of the respective treatment period
  Participants will self-report the number of days in the two week rinsing period in which they used rinses.

OTHER OUTCOMES:
Frequency (by severity) of adverse effects after sinus rinses | From the beginning of week 2 to the end of week 3 of the respective treatment period
  The frequency (by severity) of the following patient-reported adverse effects:
  * Nasal burning/pain
  * Headaches
  * Ear pain
  * Sneezing
  * Nose bleeds

CONTACTS AND LOCATIONS:
Overall Officials: Neelaysh Vukkadala, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No